CLINICAL TRIAL: NCT06320210
Title: Chicago Asthma School-Directed Child-Centered Assessment and Dissemination of Evidence
Acronym: CASCADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB19-1308
Record Dates: First submitted 2024-03-12; First posted 2024-03-20 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with asthma, parents/guardians of children with asthma, school staff (Experimental): Children will be recruited from two University of Chicago Charter elementary schools. Children with a diagnosis of asthma and their parents will be eligible for inclusion in the study and will specifically be targeted for study recruitment. Staff and administrators at each school will also be recruited through in-person, phone, and email communication, primarily through word of mouth and professional development days. UCCS teachers, staff, and administrators will also be included in the program evaluation and we will obtain appropriate consent.
  Up to 400 families with a child/children with asthma from two UCCS schools will be added to a registry database. A total of 68 children with a diagnosis of asthma and their parents will be recruited for evaluation of the multi-component program, resulting in a total of 136 children and parents. We will also recruit 24 teachers, staff, and administrators across the two schools to participate in the evaluation of the overall program.
  Interventions: Behavioral: Multicomponent program

INTERVENTIONS:
Behavioral: Multicomponent program — The intervention is a multi-component program that includes in-depth training for current school teachers/staff who are critical in asthma care, restructured processes to identify students with asthma, technological adaptations to support integrated systems for asthma care and absenteeism, strategies to enhance communication about asthma within school and between school and home, protocols for routine care (e.g., participation in gym/recess) and emergencies, and education for all students about asthma.

SUMMARY:
Research has shown that adherence to evidence-based asthma guidelines leads to improved outcomes, yet critical gaps remain in the implementation of these guidelines, particularly among minority and low-income youth. Schools represent a crucial point of intervention, as demonstrated by school-based asthma programs that have addressed individual components of the guidelines with promising results. This project aims to develop, implement, and evaluate a pragmatic, multi-component asthma program that builds upon existing targeted interventions to fully implement the asthma guidelines and integrate them in school practices to foster sustainability. The investigator seeks to understand whether this type of program will improve asthma outcomes at the child and school level.

DETAILED DESCRIPTION:
Significant health disparities persist in childhood asthma prevalence and morbidity despite existing evidence-based asthma guidelines that have been shown to improve outcomes. Schools are an integral partner in asthma management. Prior literature has outlined various targeted school-based interventions with some positive outcomes; however, these programs focus on individual components of the guidelines and take place transiently without integration into school processes for sustainability. To more comprehensively impact asthma care, schools have enacted policies to support guideline-based practices; however, implementation falls short and thus these policies have not led to effective, systemic practices. Therefore, this project aims to bridge the gap in the implementation of asthma guidelines and policies by developing and evaluating a pragmatic, multicomponent school-directed, child-centered asthma program that builds upon existing targeted interventions and is integrated in the school to foster sustainability. This innovative project contributes beyond existing school-based programs by simultaneously and pragmatically implementing multiple components of the asthma guidelines through school-wide systems and streamlined processes led by lay health workers.

A multi-level program will be put in place for all students and families within the school. Intervention components will include: in-depth training for current school staff who are critical in asthma care, restructured processes to identify students with asthma, technological adaptations to create integrated tracking systems for asthma care and absenteeism, strategies to enhance communication about asthma within school and between school and home, protocols for routine care (e.g., participation in gym/recess) and emergencies, and education for all students about asthma.

ELIGIBILITY:
Participants will be included in the study if:

1. The participant either works at, attends, or is the legal guardian of a child who attends one of the two elementary schools included in the study from the University of Chicago Charter Schools - North Kenwood Oakland and Donoghue.
2. The child participant has a diagnosis of asthma OR the parent participant is legal guardian of a child with asthma.
3. The adult stakeholder is 18 years or older.

Participants will be excluded from the study if:

1. The participant declines or is unable to provide consent/assent
2. The participant does not speak or read English
3. The participant has already enrolled in the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Asthma control | Years 1 and 2
  Childhood Asthma Control Test

SECONDARY OUTCOMES:
Missed work days in parents | Years 1 and 2
  Parent reports, logs
Asthma knowledge - parents | Years 1 and 2
  Asthma Knowledge Scale
Asthma knowledge - child | Years 1 and 2
  Asthma Knowledge Scale
Asthma quality of life - child | Years 1 and 2
  Pediatric Asthma Quality of Life Questionnaire
Caregiver quality of life | Years 1 and 2
  Pediatric Asthma Caregiver's Quality of Life Questionnaire
Asthma impact - parent | Years 1 and 2
  Parent Proxy Asthma Impact Scale
Missed school days | Years 1 and 2
  School records, parent report, logs
Healthcare utilization | Years 1 and 2
  Parent report and logs of ambulatory visits, emergency department visits, hospitalizations
Asthma impact - child | Years 1 and 2
  Pediatric Asthma Impact Scale

CONTACTS AND LOCATIONS:
Overall Officials: Anna Volerman, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Charter Schools, Chicago, Illinois, United States

REFERENCES:
- [Background] Bloom B, Jones LI, Freeman G. Summary health statistics for U.S. children: National Health Interview Survey, 2012. Vital Health Stat 10. 2013 Dec;(258):1-81. PMID 24784481
- [Background] National Surveillance of Asthma: United States, 2001-2010. Hyattsville, MD: U.S. Dept. of Health and Human Services, Centers for Disease Control and Prevention, National Center for Health Statistics; 2012.
- [Background] Centers for Disease Control and Prevention. Asthma Data, Statistics, and Surveillance. Most Recent Asthma Data. 2017.
- [Background] Centers for Disease Control and Prevention. Asthma-Related Missed School Days among Children Aged 5-17 Years.; 2015.
- [Background] Quinn K, Shalowitz MU, Berry CA, Mijanovich T, Wolf RL. Racial and ethnic disparities in diagnosed and possible undiagnosed asthma among public-school children in Chicago. Am J Public Health. 2006 Sep;96(9):1599-603. doi: 10.2105/AJPH.2005.071514. Epub 2006 Feb 28. PMID 16507720
- [Background] Akinbami LJ, Simon AE, Rossen LM. Changing Trends in Asthma Prevalence Among Children. Pediatrics. 2016 Jan;137(1):1-7. doi: 10.1542/peds.2015-2354. Epub 2015 Dec 28. PMID 26712860
- [Background] Gupta RS, Zhang X, Sharp LK, Shannon JJ, Weiss KB. Geographic variability in childhood asthma prevalence in Chicago. J Allergy Clin Immunol. 2008 Mar;121(3):639-645.e1. doi: 10.1016/j.jaci.2007.11.036. Epub 2008 Feb 4. PMID 18243285
- [Background] Illinois Department of Public Health. The Burden of Asthma in Illinois, 2000-2011. State of Illinois; 2013.
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Volerman A, Kan K, Salem E, Prachand N, Warren CM, Sighoko D, Gupta RS. Disparities persist in asthma-related emergency department visits among Chicago children. Ann Allergy Asthma Immunol. 2019 Apr;122(4):417-419.e1. doi: 10.1016/j.anai.2019.01.011. Epub 2019 Jan 24. No abstract available. PMID 30684738
- [Background] National Heart, Lung, and Blood Institute. Guidelines for the Diagnosis and Management of Asthma: Expert Panel Report 3. Washington, DC: US Department of Health and Human Services; 2007.
- [Background] National Heart, Lung, and Blood Institute. Managing Asthma: A Guide for Schools. Washington, DC: US Department of Health and Human Services; 2014.
- [Background] Asthma Management Policy. Chicago Public Schools Policy Manual; 2012.
- [Background] Cloutier MM, Hall CB, Wakefield DB, Bailit H. Use of asthma guidelines by primary care providers to reduce hospitalizations and emergency department visits in poor, minority, urban children. J Pediatr. 2005 May;146(5):591-7. doi: 10.1016/j.jpeds.2004.12.017. PMID 15870660
- [Background] Grant EN, Malone A, Lyttle CS, Weiss KB. Asthma morbidity and treatment in the Chicago metropolitan area: one decade after national guidelines. Ann Allergy Asthma Immunol. 2005 Jul;95(1):19-25. doi: 10.1016/S1081-1206(10)61183-0. PMID 16095137
- [Background] Mattke S, Martorell F, Sharma P, Malveaux F, Lurie N. Quality of care for childhood asthma: estimating impact and implications. Pediatrics. 2009 Mar;123 Suppl 3:S199-204. doi: 10.1542/peds.2008-2233K. PMID 19221164
- [Background] Wolf RL, Berry CA, O'Connor T, Coover L. Validation of the Brief Pediatric Asthma Screen. Chest. 1999 Oct;116(4 Suppl 1):224S-228S. doi: 10.1378/chest.116.suppl_2.224s. PMID 10532498
- [Background] Wolf RL, Berry CA, Quinn K. Development and validation of a brief pediatric screen for asthma and allergies among children. Ann Allergy Asthma Immunol. 2003 May;90(5):500-7. doi: 10.1016/S1081-1206(10)61843-1. PMID 12775131
- [Background] Redline S, Gruchalla RS, Wolf RL, Yawn BP, Cartar L, Gan V, Nelson P, Wollan P. Development and validation of school-based asthma and allergy screening questionnaires in a 4-city study. Ann Allergy Asthma Immunol. 2004 Jul;93(1):36-48. doi: 10.1016/S1081-1206(10)61445-7. PMID 15281470
- [Background] Gupta RS, Ballesteros J, Springston EE, Smith B, Martin M, Wang E, Damitz M. The state of pediatric asthma in Chicago's Humboldt Park: a community-based study in two local elementary schools. BMC Pediatr. 2010 Jun 24;10:45. doi: 10.1186/1471-2431-10-45. PMID 20576150
- [Background] Gupta RS, Lau CH, Warren CM, Lelchuk A, Alencar A, Springston EE, Holl JL. The impact of student-directed videos on community asthma knowledge. J Community Health. 2013 Jun;38(3):463-70. doi: 10.1007/s10900-012-9630-4. PMID 23184318
- [Background] Christiansen SC, Martin SB, Schleicher NC, Koziol JA, Mathews KP, Zuraw BL. Evaluation of a school-based asthma education program for inner-city children. J Allergy Clin Immunol. 1997 Nov;100(5):613-7. doi: 10.1016/s0091-6749(97)70164-7. PMID 9389290
- [Background] Gerald LB, McClure LA, Mangan JM, Harrington KF, Gibson L, Erwin S, Atchison J, Grad R. Increasing adherence to inhaled steroid therapy among schoolchildren: randomized, controlled trial of school-based supervised asthma therapy. Pediatrics. 2009 Feb;123(2):466-74. doi: 10.1542/peds.2008-0499. PMID 19171611
- [Background] Halterman JS, Riekert K, Bayer A, Fagnano M, Tremblay P, Blaakman S, Borrelli B. A pilot study to enhance preventive asthma care among urban adolescents with asthma. J Asthma. 2011 Jun;48(5):523-30. doi: 10.3109/02770903.2011.576741. PMID 21599562
- [Background] Anderson ME, Freas MR, Wallace AS, Kempe A, Gelfand EW, Liu AH. Successful school-based intervention for inner-city children with persistent asthma. J Asthma. 2004 Jun;41(4):445-53. doi: 10.1081/jas-120033987. PMID 15281330
- [Background] Halterman JS, Szilagyi PG, Fisher SG, Fagnano M, Tremblay P, Conn KM, Wang H, Borrelli B. Randomized controlled trial to improve care for urban children with asthma: results of the School-Based Asthma Therapy trial. Arch Pediatr Adolesc Med. 2011 Mar;165(3):262-8. doi: 10.1001/archpediatrics.2011.1. PMID 21383275
- [Background] Harris K, Kneale D, Lasserson TJ, McDonald VM, Grigg J, Thomas J. School-based self-management interventions for asthma in children and adolescents: a mixed methods systematic review. Cochrane Database Syst Rev. 2019 Jan 28;1(1):CD011651. doi: 10.1002/14651858.CD011651.pub2. PMID 30687940
- [Background] Bruzzese JM, Evans D, Kattan M. School-based asthma programs. J Allergy Clin Immunol. 2009 Aug;124(2):195-200. doi: 10.1016/j.jaci.2009.05.040. Epub 2009 Jul 16. PMID 19615728
- [Background] Coffman JM, Cabana MD, Yelin EH. Do school-based asthma education programs improve self-management and health outcomes? Pediatrics. 2009 Aug;124(2):729-42. doi: 10.1542/peds.2008-2085. Epub 2009 Jul 27. PMID 19651589
- [Background] Coffman JM, Cabana MD, Halpin HA, Yelin EH. Effects of asthma education on children's use of acute care services: a meta-analysis. Pediatrics. 2008 Mar;121(3):575-86. doi: 10.1542/peds.2007-0113. PMID 18310208
- [Background] Wheeler LS, Merkle SL, Gerald LB, Taggart VS. Managing asthma in schools: lessons learned and recommendations. J Sch Health. 2006 Aug;76(6):340-4. doi: 10.1111/j.1746-1561.2006.00125.x. No abstract available. PMID 16918868
- [Background] Wheeler L, Buckley R, Gerald LB, Merkle S, Morrison TA. Working With Schools to Improve Pediatric Asthma Management. Pediatric Asthma, Allergy & Immunology. 2009;22(4):197-208.
- [Background] Wolf FM, Guevara JP, Grum CM, Clark NM, Cates CJ. Educational interventions for asthma in children. Cochrane Database Syst Rev. 2003;2002(1):CD000326. doi: 10.1002/14651858.CD000326. PMID 12535395
- [Background] Volerman A, Chin MH, Press VG. Solutions for Asthma Disparities. Pediatrics. 2017 Mar;139(3):e20162546. doi: 10.1542/peds.2016-2546. Epub 2017 Feb 22. No abstract available. PMID 28228500
- [Background] Volerman A, Ignoffo S, Hull A, McArthur Hanshaw S, Taylor S, Vela M, Press VG. Identification of students with asthma in Chicago schools: Missing the mark. Ann Allergy Asthma Immunol. 2017 Jun;118(6):739-740. doi: 10.1016/j.anai.2017.04.004. Epub 2017 May 4. No abstract available. PMID 28479193
- [Background] Volerman A, Dennin M, Vela M, Ignoffo S, Press VG. A qualitative study of parent perspectives on barriers, facilitators and expectations for school asthma care among urban, African-American children. J Asthma. 2019 Oct;56(10):1099-1109. doi: 10.1080/02770903.2018.1520861. Epub 2018 Oct 4. PMID 30285497
- [Background] Naman J, Press VG, Vaughn D, Hull A, Erwin K, Volerman A. Student perspectives on asthma management in schools: a mixed-methods study examining experiences, facilitators, and barriers to care. J Asthma. 2019 Dec;56(12):1294-1305. doi: 10.1080/02770903.2018.1534968. Epub 2018 Oct 30. PMID 30376385